CLINICAL TRIAL: NCT02395692
Title: Phase II Study of TRC102 in Combination With Temozolomide for Recurrent Glioblastoma
Brief Title: Methoxyamine and Temozolomide in Treating Patients With Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pre-specified response criteria not met to proceed to next stage of study.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00356; NCI-2015-00356 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1402 (Other: Adult Brain Tumor Consortium); ABTC-1402 (Other: Adult Brain Tumor Consortium); ABTC 1402 (Other: Adult Brain Tumor Consortium); ABTC-1402 (Other: CTEP); UM1CA137443 (NIH)
Record Dates: First submitted 2015-03-23; First posted 2015-03-24 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Adult Brain Glioblastoma
MeSH Terms: interventions — Therapeutics; methoxyamine; Temozolomide

ARMS (1):
- Treatment (methoxyamine, temozolomide) (Experimental): Patients receive methoxyamine PO QD and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Treatment; Drug: Methoxyamine; Drug: Temozolomide

INTERVENTIONS:
Other: Treatment — Correlative studies
Drug: Methoxyamine — Given PO
  Other Names: TRC102
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase II trial studies how well methoxyamine works when added to standard temozolomide in treating patients with glioblastoma that has come back. Drugs used in chemotherapy, such as methoxyamine and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the efficacy of TRC102 (methoxyamine) and temozolomide, as measured by response rate, in bevacizumab naïve glioblastoma. (Arm I) II. To estimate the efficacy of TRC102 and temozolomide, as measured by response rate, in bevacizumab refractory glioblastoma. (Arm II)

SECONDARY OBJECTIVES:

I. Evaluate the toxicities of oral TRC102 and temozolomide in this patient population.

II. Estimate the efficacy of TRC102 and temozolomide, as measured by progression-free survival, progression-free survival at 6 months and overall survival, in bevacizumab naïve glioblastoma.

III. Estimate the efficacy of TRC102 and temozolomide, as measured by progression-free survival in bevacizumab refractory glioblastoma.

TERTIARY OBJECTIVES:

I. Assess the tissue correlates of N-methylpurine-deoxyribonucleic acid (DNA) glycosylase (MPG), topoisomerase II-alpha (topo II a), and O-6-methylguanine-DNA methyltransferase (MGMT) status, with response, progression-free survival (PFS), and overall survival.

OUTLINE:

Patients receive methoxyamine orally (PO) once daily (QD) and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, every 2 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed glioblastoma that is progressive or recurrent following radiation therapy and temozolomide
* Tumor MGMT methylation status must be available; results of routinely used methods for MGMT methylation testing (e.g. methylation-specific polymerase chain reaction [MSPCR ] or quantitative polymerase chain reaction [PCR]) are acceptable
* Arm 1 patients must have measurable (defined by at least 1 cm x 1 cm) contrast-enhancing disease by magnetic resonance imaging (MRI) imaging within 21 days of starting treatment
* Patients must be able to undergo MRI of the brain with gadolinium; patients must be maintained on a stable or decreasing dose of corticosteroid regimen (no increase for 5 days) prior to this baseline MRI
* Arm 1 patients must be in first recurrence of glioblastoma following radiation therapy and temozolomide
* Arm 2 patients may have an unlimited number of prior therapy regimens but may not have received prior antiangiogenesis therapy except for bevacizumab (patients may not have received aflibercept, ramucirumab, cediranib, cabozantinib, or XL184)
* Arm 1 patients must have not received bevacizumab previously
* Arm 2 patients must have progressed/recurred on bevacizumab as the most recent regimen; patients on arm 2 should continue on bevacizumab as clinically necessary to control brain edema
* Patients must have a tumor tissue form indicating availability of archived tissue from initial resection at diagnosis of glioblastoma completed and signed by a pathologist; availability of tissue is not a requirement for study participation
* Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., erlotinib, hydroxychloroquine, etc.)
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 4 x institutional upper limit of normal
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Activated partial thromboplastin time (APTT) or partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
* Patients must be able to provide written informed consent
* Women of childbearing potential must have a negative serum pregnancy test prior to study start; women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and through 30 days after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and through 30 days after the last dose of study drug
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
* Patients must be able to swallow capsules

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible
* Patient must not have known sensitivity to TRC102 or any formulation excipients
* Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol; patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs; patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of TRC102
* Patients must not be on any anticoagulation
* Patient must not have prior gastrointestinal (GI) surgery or GI disease that might interfere with the absorption of TRC102
* Patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to prior therapy are ineligible
* Patients must not have active brain metastases from a systemic solid tumor
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with TRC102
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, Principal Investigator — National Cancer Institute (NCI)
Locations (12):
- United States (12):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Adult Brain Tumor Consortium, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Henry Ford Cancer Institute¿Downriver, Brownstown, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject withdrew before start of study
Groups:
- Arm1 Methoxyamine &Temozolomide (Bevacizumab-naïve): Patients receive methoxyamine PO QD and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Bevacizumab-naive
  Laboratory Biomarker Analysis: Correlative studies
  Methoxyamine: Given PO
  Temozolomide: Given PO
- Arm2 Methoxyamine & Temozolomide (Bevacizumab-refractory): Patients receive methoxyamine PO QD and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Bevacizumab-refractory
  Laboratory Biomarker Analysis: Correlative studies
  Methoxyamine: Given PO
  Temozolomide: Given PO
Period: Overall Study
Arm/Group | Arm1 Methoxyamine &Temozolomide (Bevacizumab-naïve) | Arm2 Methoxyamine & Temozolomide (Bevacizumab-refractory)
Started | 19 | 0
Completed | 19 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Methoxyamine, Temozolomide): Patients receive methoxyamine PO QD and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Methoxyamine: Given PO
  Temozolomide: Given PO
Arm/Group | Treatment (Methoxyamine, Temozolomide)
Number analyzed (Participants) | 19
Age, Customized [Median (Full Range); unit: years] | 60 [48 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19
Karnofsky Performance Score (KPS) [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 80 [70 to 90]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response as Assessed by Response Assessment in Neuro-Oncology (RANO) Criteria (Arm 1 and Arm 2)
Description: To test the hypothesis that the combination treatment of temozolomide and methoxyamine will achieve 30% radiographic response rate (partial response + complete response) in patients with first recurrence of glioblastoma.
  Per Response Assessment in Neuro-Oncology (RANO) Criteria: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to at least 2 years
Population: This was a 2 stage design study. if there were less than 2 responders in first 19 subjects, study would terminate and Arm2 would not accrue any subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Arm1 Methoxyamine&Temozolomide (Bevacizumab-naïve): Patients receive methoxyamine PO QD and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. (Bevacizumab-naïve)
  Laboratory Biomarker Analysis: Correlative studies
  Methoxyamine: Given PO
  Temozolomide: Given PO
- Arm2 Methoxyamine&Temozolomide (Bevacizumab-refractory): Patients receive methoxyamine PO QD and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Bevacizumab-refractory
  Laboratory Biomarker Analysis: Correlative studies
  Methoxyamine: Given PO
  Temozolomide: Given PO
Arm/Group | Arm1 Methoxyamine&Temozolomide (Bevacizumab-naïve) | Arm2 Methoxyamine&Temozolomide (Bevacizumab-refractory)
Number analyzed (Participants) | 19 | 0
Participants | 0 |

2. Secondary Outcome: Toxicity as Assessed by Number of Participants Who Experienced Adverse Events
Description: Number of participants who experience adverse events graded 3 or higher as defined by National Cancer Institute CTCAE v4.0.
Time Frame: Up to 30 days following the last dose of study drug
Population: Patients diagnosed with glioblastoma
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Methoxyamine, Temozolomide): Patients receive methoxyamine PO QD and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Treatment (methoxyamine, temozolomide): Correlative studies
  Methoxyamine: Given PO
  Temozolomide: Given PO
Arm/Group | Treatment (Methoxyamine, Temozolomide)
Number analyzed (Participants) | 19
Participants | 19

3. Secondary Outcome: Progression-free Survival
Description: Will be analyzed using standard descriptive statistical methods. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to at least 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Methoxyamine, Temozolomide)
Number analyzed (Participants) | 19
months | 2 [1.8 to 3.6]

4. Secondary Outcome: Progression-free Survival at 6 Months
Description: Will be analyzed using standard descriptive statistical methods.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Methoxyamine, Temozolomide)
Number analyzed (Participants) | 19
Participants | 2

5. Secondary Outcome: Overall Survival
Description: Will be analyzed using standard descriptive statistical methods.
Time Frame: Up to at least 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Methoxyamine, Temozolomide)
Number analyzed (Participants) | 19
months | 11 [8 to 18]

6. Other Pre Specified Outcome: MPG, Topo II-alpha, and MGMT Levels in Tissue Samples
Description: MPG, topo II-alpha, and MGMT levels will be correlated with response, PFS, and overall survival. Will be analyzed using standard descriptive statistical methods.
Time Frame: Baseline
Population: Data was not collected to assess this outcome measure.
Arm/Group | Treatment (Methoxyamine, Temozolomide)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 and 30 days after the last dose of the study drug
Arm/Group | Treatment (Methoxyamine, Temozolomide)
All-Cause Mortality (participants affected / at risk) | 9/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 18/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Methoxyamine, Temozolomide) (N=19)
Alanine Aminotransferase increased (Investigations) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 17 (42)
anorexia (Metabolism and nutrition disorders) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Blood bilirubin increased (Investigations) | 9 (9)
Constipation (Gastrointestinal disorders) | 9 (10)
diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Dysphasia (Nervous system disorders) | 2 (2)
fatigue (General disorders) | 7 (11)
Fever (General disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (5)
Lymphocyte count decreased (Investigations) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (8)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 4 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
White blood cell decreased (Investigations) | 10 (21)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Investigations - Other, TRIGLYCERIDES HIGH (Investigations) | 1 (1) — TRIGLYCERIDES HIGH Investigations - Other, specify; 10022891
Alkaline phosphatase increased (Investigations) | 1 (1)
INCREASED BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 (1)
COLON POLYP (Gastrointestinal disorders) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — UPPER BACK, LEFT UPPER ARM, LEFT GROIN
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders - Other, EXTREMELY HOT SENSATION (Nervous system disorders) | 1 (1) — EXTREMELY HOT SENSATION
Nervous system disorders - Other, Vasogenic Edema (Nervous system disorders) | 1 (1) — Vasogenic Edema
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, SORE IN GROIN AREA (Skin and subcutaneous tissue disorders) | 1 (1) — SORE IN GROIN AREA
Stroke (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight Gain (Investigations) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
n for this study 31 subjects w/ a 2 stage design. 19 subjects were treated in stage one with TRC102 and TMZ in recurrent GBM. If no more than 2 responses were observed among the initial 19 patients the study would be terminated and declared negative

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT02395692/Prot_SAP_000.pdf